CLINICAL TRIAL: NCT03980938
Title: A Double-Blind, Placebo-Controlled Two-Period 10-Week Treatment Within-Subject Crossover Study Of Cognitive Effects Of Neflamapimod in Early-Stage Huntington Disease (HD)
Brief Title: Within Subject Crossover Study of Cognitive Effects of Neflamapimod in Early-Stage Huntington Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the long delay because of COVID-19 and results from another study suggesting a higher dose may be more beneficial, EIP Pharma decided on October 15th, 2020, to end the trial prematurely.
Sponsor: EIP Pharma Inc (Industry)
Collaborators: Voisin Consulting, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIP19-NFD-401
Record Dates: First submitted 2019-06-07; First posted 2019-06-10 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — VX-745

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- neflamapimod first (Experimental): neflamapimod in Treatment Period 1, placebo in Treatment Period 2
  neflamapimod: 40 mg neflamapimod hard gelatin capsules, taken twice daily with food.
  Placebo: hard gelatin capsules containing excipients only, weight- and size-matched; taken twice daily with food.
  Interventions: Drug: neflamapimod; Other: Placebo
- placebo first (Placebo Comparator): placebo in Treatment Period 1, neflamapimod in Treatment Period 2
  Placebo: hard gelatin capsules containing excipients only, weight- and size-matched; taken twice daily with food.
  neflamapimod: 40 mg neflamapimod hard gelatin capsules, taken twice daily with food.
  Interventions: Drug: neflamapimod; Other: Placebo

INTERVENTIONS:
Drug: neflamapimod — 40 mg neflamapimod capsule
  Other Names: VX-745
Other: Placebo — matching placebo capsule

SUMMARY:
This is a double-blind, placebo-controlled 2-period 10-week treatment within-subject crossover study of neflamapimod in early-stage Huntington disease (HD). The primary objective is to determine whether neflamapimod can reverse hippocampal dysfunction in patients with early-stage HD, as assessed by the virtual water-maze-test for evaluating spatial learning and selected tests on the Cambridge Neuropsychological Test Automated Battery (CANTAB).

DETAILED DESCRIPTION:
The study was designed as within-subject crossover study. However, due to the Covid19 lockdowns and restrictions on clinical research, and only one subject entered the second crossover period. As a result, the baseline and outcomes are reported by the actual treatment received in the subjects during what would have been the first treatment period, i.e. placebo or neflamapimod treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 30 to 70 years, inclusive.
2. Willing and able to provide informed consent.
3. Must have genetically confirmed HD and identified cognitive deficits:

   1. Stage 1, as defined by Unified Huntington's Disease Rating Scale (UHDRS) Total Functional Capacity (TFC) score >10, and,
   2. CANTAB Paired Associate Learning Total Adjusted Error Score of >16.
4. Normal or corrected eye sight and auditory abilities, sufficient to perform all aspects of the cognitive and functional assessments.
5. No history of learning difficulties that may interfere with the subject's ability to complete the cognitive tests.

Exclusion Criteria:

1. A profile of impairment that is not consistent with HD.
2. Diagnosis of any other ongoing central nervous system condition other than HD, including, but not limited to, vascular dementia, dementia with Lewy bodies, and Parkinson's disease.
3. Suicidality, defined as active suicidal thoughts within 6 months before Screening or at Baseline, defined as answering yes to items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS), or history of suicide attempt in previous 2 years, or, in the Investigator's opinion, at serious risk of suicide.
4. Ongoing major and active psychiatric disorder, moderate to severe depressive symptoms, and or other concurrent medical condition that, in the opinion of the Investigator, might compromise safety and/or compliance with study requirements.
5. Diagnosis of alcohol or drug abuse within the previous 2 years.
6. Poorly controlled clinically significant medical illness, such as hypertension (blood pressure >180 mmHg systolic or 100 mmHg diastolic); myocardial infarction within 6 months; uncompensated congestive heart failure or other significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude treatment with p38 mitogen activated protein (MAP) kinase inhibitor and/or assessment of drug safety and efficacy.
7. Anemia with a hemoglobin ≤10 g/dL, clinically significant thyroid function abnormality, electrolyte abnormalities.
8. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 × the upper limit of normal (ULN), total bilirubin >1.5 × ULN, and/or International Normalized Ratio (INR) >1.5.
9. Known human immunodeficiency virus; or active hepatitis B or hepatitis C virus infection; evidence of active or latent tuberculosis.
10. Subject participated in a study of an investigational drug less than 3 months or 5 half-lives of an investigational drug, whichever is longer, before enrollment in this study.
11. History of previous neurosurgery to the brain.
12. Female subjects who are pregnant or breast-feeding.
13. Male subjects with female partners of child-bearing potential who are unwilling or unable to adhere to contraception requirements specified in the protocol (see Section 5.8).
14. Female subjects who have not reached menopause or have not had a hysterectomy or bilateral oophorectomy/salpingo-oophorectomy and are not willing or unable to adhere to contraceptive requirements specified in the protocol (see Section 5.8).
15. Requires concomitant use of cytochrome P450 (CYP) 3A4 inhibitors or anti-tumor necrosis factor-alpha therapies during study participation.
16. Known allergy to any ingredient of the trial medication or placebo.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Alam, MD, Study Director — EIP Pharma
Locations (1):
- John Van Geest Centre for Brain Repair, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tormahlen NM, Martorelli M, Kuhn A, Maier F, Guezguez J, Burnet M, Albrecht W, Laufer SA, Koch P. Design and Synthesis of Highly Selective Brain Penetrant p38alpha Mitogen-Activated Protein Kinase Inhibitors. J Med Chem. 2022 Jan 27;65(2):1225-1242. doi: 10.1021/acs.jmedchem.0c01773. Epub 2021 May 11. PMID 33974419

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Neflamapimod First | Placebo First
Started | 7 | 8
Completed | 6 | 7
Not Completed | 1 | 1
Not completed — Study Terminated | 1 | 1
Period: Treatment Period 2
Arm/Group | Neflamapimod First | Placebo First
Started (The study was halted in March 2020 due to COVID-19 pandemic and eventually terminated without resuming any study activities. At this time 5 participants had started Treatment Period 2. 2 participants were in Treatment Period 1 and 8 participants were in the Washout Period, thus 10 participants never started Treatment Period 2.) | 3 | 2
Completed | 1 (One participant completed the study remotely. On-site visits were no longer permitted due to COVID-19 pandemic. Visits were conducted remotely for Weeks 8 and 10 of Treatment Period 2, and the follow-up visit.) | 0
Not Completed | 2 | 2
Not completed — Study Terminated | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neflamapimod First | Placebo First | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12.26) | 54.5 (9.68) | 52.87 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 8 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 8 | 15
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 26.3 (5.4) | 27.61 (6.15) | 27 (5.65)

OUTCOME MEASURES:

1. Primary Outcome: Change in Latency During the Learning Phase of Virtual Morris Water Maze Test (vMWM)
Description: Change from baseline of latency during the learning phase of vMWM (hidden platform training) in the neflamapimod first group compared to placebo first group
Time Frame: Baseline and 10 Weeks
Population: Participants who had analyzable results at Baseline and Week 10 of Treatment Period 1 (13 participants)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Neflamapimod First | Placebo First
Number analyzed (Participants) | 6 | 7
seconds | -6.92 (3.814) | -14.05 (12.680)

ADVERSE EVENTS:
Time Frame: Up to 37 weeks. AEs occurring from when the subject signed the ICF until up to 30 days after the last dose were collected. Any AEs occurring before the start of treatment (i.e., before the first dose of the investigational product) were recorded in the medical history.
Description: Any sign, symptom, or disease present before starting the treatment period were only considered AEs if they worsen after starting the treatment period.
  All-Cause Mortality was not monitored/assessed.
Arm/Group | Neflamapimod First | Placebo First
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 4/7 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neflamapimod First (N=7) | Placebo First (N=8)
Common Cold (Infections and infestations) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sores (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Increased Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due COVID-19 pandemic all clinical research in the UK was halted in March 2020. Sponsor ultimately elected to terminate the study on 15 October 2020. As only one subject completed both periods of the crossover, the only efficacy analyses compared outcomes in subjects receiving neflamapimod (N=7) during Treatment period 1 to those receiving placebo during that period (N=8); i.e., an inter-subject group comparison, rather than the within-subject comparison for which the study was powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT03980938/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT03980938/SAP_001.pdf